CLINICAL TRIAL: NCT02363959
Title: Hyperbaric Oxygen Therapy for Lung Transplantation-Associated Pseudomembranes and Central Airway Stenosis
Brief Title: Hyperbaric Oxygen Therapy for Lung Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00055849
Record Dates: First submitted 2015-02-10; First posted 2015-02-16 (Estimated); Results first posted 2019-10-17 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Disorder Related to Lung Transplantation; Central Airway Stenosis; Airway Exudative Plaques; Airway Complications Post-Lung Transplantation
Keywords: Hyperbaric Oxygen; Lung Transplantation; Central Airway Stenosis; Airway Exudative Plaques; Hyperbaric Oxygen Therapy; Post-Lung Transplantation; Airway Ischemia; Endobronchial Biopsy; Bronchoscopy
MeSH Terms: interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hyperbaric Oxygen, Airway Biopsy (Experimental): The hyperbaric oxygen therapy (HBOT) will be performed with the standard HBOT protocol used at Duke for the treatment of compromised grafts and flaps. This is 2 hours of breathing >99% medical grade oxygen inside an air-pressurized chamber at atmospheric pressure of 2 (2 ATA) once a day for 20 sessions. These sessions will be scheduled 3-5 times per week, depending on the availability of the patient and the hyperbaric medicine physician.
  During standard bronchoscopies, an endobronchial biopsy of the airway epithelium will be performed. Biopsy will add roughly 3 minutes total to each procedure.
  Interventions: Drug: Hyperbaric Oxygen Therapy; Procedure: Endobronchial Biopsy of Airway Epithelium
- No Hyperbaric Oxygen, Airway Biopsy (Other): No hyperbaric oxygen therapy administered, but lung biopsy still completed during standard post-lung transplant bronchoscopies. An endobronchial biopsy of the airway epithelium will be performed. Biopsy will add roughly 3 minutes total to each procedure.
  Interventions: Procedure: Endobronchial Biopsy of Airway Epithelium

INTERVENTIONS:
Drug: Hyperbaric Oxygen Therapy — 2 hours of breathing >99% medical grade oxygen inside an air-pressurized chamber at 2 ATA once a day for 20 sessions. These sessions will be scheduled 3-5 times per week, depending on the availability of the patient and the hyperbaric medicine physician.
  Other Names: HBOT; Hyperbaric Oxygen
  Arms: Hyperbaric Oxygen, Airway Biopsy
Procedure: Endobronchial Biopsy of Airway Epithelium — During standard post-transplantation bronchoscopies, participants in this study will undergo an endobronchial biopsy of the airway epithelium for each donor lung.
  Other Names: Airway Biopsy

SUMMARY:
The objective of this study is to evaluate the effect of hyperbaric oxygen therapy (HBOT) on airway complications in post-lung transplant recipients with evidence of restricted levels of blood and oxygen in the airway tissue. Study subjects with extensive airway tissue damage in the early post-transplant period will be randomized to HBOT or usual care and followed clinically for 12 months following randomization. The investigators hypothesize that HBOT will decrease the number of airway complications in the treated subjects.

DETAILED DESCRIPTION:
Hyperbaric oxygen therapy (HBOT) will be performed with the standard HBOT protocol used at Duke for the treatment of compromised grafts and flaps. This is 2 hours of breathing >99% medical grade oxygen inside an air-pressurized chamber at atmospheric pressure of 2 once a day for 20 sessions. These sessions will be scheduled 3-5 times per week, depending on the availability of the patient and the hyperbaric medicine physician. The HBOT procedure used for this study will be identical to that used for clinical practice in the Duke University Health System Center for Hyperbaric Medicine and Environmental Physiology, including the oxygen that is used in the chamber. Patients will receive treatment through the regular clinical hyperbaric service. These are routine, not special, treatment sessions and they will receive them alongside other Duke University Medical Center patients being treated for other reasons. The medical grade oxygen used is a part of the Duke University Health System Center for Hyperbaric Medicine and Environmental Physiology hyperbaric chamber system.

While the patients randomized to receive usual care will not undergo HBOT, both study groups will receive standard serial bronchoscopies for airway clearance and for the collection of bronchoalveolar lavage fluid for culture data, due to the high rate of infection in lung transplant patients. All subjects will undergo the standard surveillance bronchoscopies every 3 to 4 weeks (x3) for clearance of the exudate from the airway, as well as monitoring progression of the airway abnormalities. As participants in this study, an, endobronchial biopsy of the airway epithelium will be performed at the main carina to collect a sample of recipient epithelium as well as at the first subcarina for each donor lung. Three samples will be collected from each of the biopsy sites. These samples are small (1 to 2 mm) and are thought to have a minimal clinical risk of minor bleeding associated with the procedure. Biopsy will add roughly 3 minutes total to each procedure.

ELIGIBILITY:
Inclusion Criteria:

* Post-lung transplant patient
* Extensive exudative plaques at 1 month bronchoscopy
* No sign of airway improvement, or showing worsening of plaques at follow-up bronchoscopy 2-3 weeks after 1 month bronchoscopy.

Exclusion Criteria:

* Use of mechanical ventilation with fraction of inspired oxygen(FiO2) greater than 40%
* Use of extracorporeal membrane oxygenation
* Use of inhaled nitric oxide
* Presence of pneumothorax
* Pregnancy
* Inability to provide informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Shofer, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Kraft BD, Mahmood K, Harlan NP, Hartwig MG, Snyder LD, Suliman HB, Shofer SL. Hyperbaric oxygen therapy to prevent central airway stenosis after lung transplantation. J Heart Lung Transplant. 2021 Apr;40(4):269-278. doi: 10.1016/j.healun.2021.01.008. Epub 2021 Jan 15. PMID 33518452

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hyperbaric Oxygen, Airway Biopsy | No Hyperbaric Oxygen, Airway Biopsy
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0
Not completed — Medical instability | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hyperbaric Oxygen, Airway Biopsy | No Hyperbaric Oxygen, Airway Biopsy | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.65 (14.80) | 52.07 (18.76) | 52.86 (18.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Subjects Needing Airway Stent Placement as Determined by Transbronchial Lung Biopsy.
Description: Airways with stenosis refractory to serial balloon dilation x 3, or at risk for acute obstruction due to stenosis were treated with airway stents.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen, Airway Biopsy | No Hyperbaric Oxygen, Airway Biopsy
Number analyzed (Participants) | 10 | 10
Participants | 4 | 4
Statistical Analysis 1: Comparison: Hyperbaric Oxygen, Airway Biopsy vs No Hyperbaric Oxygen, Airway Biopsy; Test type: Other; p = 1, Fisher Exact; Odds Ratio (OR) = 1

2. Primary Outcome: Number of Subjects Experiencing Acute Cellular Rejection as Determined by Transbronchial Lung Biopsy
Description: Pathologic specimens will be examined for the presence of acute cellular rejection.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen, Airway Biopsy | No Hyperbaric Oxygen, Airway Biopsy
Number analyzed (Participants) | 10 | 10
Participants | 4 | 7
Statistical Analysis 1: Comparison: Hyperbaric Oxygen, Airway Biopsy vs No Hyperbaric Oxygen, Airway Biopsy; Test type: Other; p = 0.39, Fisher Exact

3. Secondary Outcome: Number of Subjects With Development of Clinically Significant Airway Stenosis
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen, Airway Biopsy | No Hyperbaric Oxygen, Airway Biopsy
Number analyzed (Participants) | 10 | 10
Participants | 5 | 4
Statistical Analysis 1: Comparison: Hyperbaric Oxygen, Airway Biopsy vs No Hyperbaric Oxygen, Airway Biopsy; Test type: Other; p = 1, Fisher Exact

4. Secondary Outcome: Number of Subjects Receiving Balloon Bronchoplasty for Management of Stenosis
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen, Airway Biopsy | No Hyperbaric Oxygen, Airway Biopsy
Number analyzed (Participants) | 10 | 10
Participants | 5 | 4
Statistical Analysis 1: Comparison: Hyperbaric Oxygen, Airway Biopsy vs No Hyperbaric Oxygen, Airway Biopsy; Test type: Other; p = 1, Fisher Exact

5. Secondary Outcome: Number of Subjects With Development of Clinically Significant Lung Infection
Description: As defined by initiation of antimicrobials to treat the suspected organism.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen, Airway Biopsy | No Hyperbaric Oxygen, Airway Biopsy
Number analyzed (Participants) | 10 | 10
Participants | 8 | 7
Statistical Analysis 1: Comparison: Hyperbaric Oxygen, Airway Biopsy vs No Hyperbaric Oxygen, Airway Biopsy; Test type: Other; p = 1, Fisher Exact

6. Secondary Outcome: Number of Subjects With Development of Bronchitis Obliterans Syndrome
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen, Airway Biopsy | No Hyperbaric Oxygen, Airway Biopsy
Number analyzed (Participants) | 10 | 10
Participants | 0 | 1
Statistical Analysis 1: Comparison: Hyperbaric Oxygen, Airway Biopsy vs No Hyperbaric Oxygen, Airway Biopsy; Test type: Other; p = 1, Fisher Exact

7. Other Pre Specified Outcome: Bronchial Epithelial Gene Expression
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Hyperbaric Oxygen, Airway Biopsy | No Hyperbaric Oxygen, Airway Biopsy
All-Cause Mortality (participants affected / at risk) | 1/10 | 1/10
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hyperbaric Oxygen, Airway Biopsy (N=10) | No Hyperbaric Oxygen, Airway Biopsy (N=10)
Repeat bronchoscopy due to bleeding during biopsy (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT02363959/Prot_SAP_000.pdf